CLINICAL TRIAL: NCT07123779
Title: Phase Ib, Multicenter, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study Assessing the Pharmacokinetics, Safety, Pharmacodynamics, and Efficacy of HS235 in Obese Patients With Pulmonary Hypertension and HFpEF
Brief Title: Study of HS235 in Obese Patients With Pulmonary Hypertension and Heart Failure With Preserved Ejection Fraction (HFpEF)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: 35Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS235-003
Record Dates: First submitted 2025-08-08; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Pulmonary Hypertension; Heart Failure With Preserved Ejection Fraction
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blinded, Placebo controlled
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Investigational Product (Experimental): HS235 Subcutaneous Injection
  Interventions: Biological: HS235
- Placebo (Placebo Comparator): Subcutaneous Injection
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: HS235 — Subcutaneous Injection
  Arms: Investigational Product
Other: Placebo — Subcutaneous Injection
  Arms: Placebo

SUMMARY:
Study of HS235 in Obese Patients with Pulmonary Hypertension and Heart Failure with Preserved Ejection Fraction Utilizing Ambulatory Pulmonary Artery Pressure Monitoring

DETAILED DESCRIPTION:
A Phase Ib, Multicenter, Double-Blind, Placebo-Controlled, Multiple Ascending Dose (MAD) Study Assessing the Pharmacokinetics, Safety, Pharmacodynamics, and Efficacy of HS235 in Obese Patients with Pulmonary Hypertension and Heart Failure with Preserved Ejection Fraction Utilizing Ambulatory Pulmonary Artery Pressure Monitoring

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible to be included in the study only if they meet at least all the following criteria:

1. Male or female, ≥ 18 years of age.
2. Ambulatory pulmonary artery pressure (PAP) monitoring (e.g. CardioMEMS™ HF System or Cordella™ HF System) implanted in the course of standard of care at least 90 days before Screening with mean pulmonary artery pressure (mPAP) ≥ 25 mmHg and diastolic pulmonary artery pressure(dPAP) ≥ 15 mmHg as averaged over the last 2 weeks prior to Randomization.
3. Established diagnosis of HFpEF with left ventricular ejection fraction (LVEF) ≥ 45 % as measured by echocardiography during Screening.
4. New York Heart Association (NYHA) class II or III heart failure symptoms.
5. Stable diuretic regimen during the screening period.
6. Kansas City Cardiomyopathy Questionnaire-Clinical Summary Score (KCCQ-CSS) < 90 at screening.
7. 6-minute walking distance (6MWD) ≥ 100 m at screening.
8. Body mass index ≥ 30 to ≤ 50 kg/m2 and Body weight ≤140 kg.
9. Ability to adhere to study visit schedule and understand and comply with all protocol requirements.

Exclusion Criteria:

1. Hospitalization for any worsening medical condition or major surgery within 4 weeks prior to screening.
2. Occurrence of an acute coronary syndrome, percutaneous coronary intervention, or cardiac surgery within 90 days prior to Screening.
3. Implantation of a cardiac resynchronization therapy (CRT) device within 90 days before screening.
4. Planned cardiovascular revascularization or planned implantation of CRT device.
5. History of heart transplant or on heart transplant list.
6. History of serious or life-threatening cardiac arrhythmia within 90 days prior to screening.
7. Systemic hypotension or uncontrolled systemic hypertension.
8. History of Pericardial constriction or hypertrophic cardiomyopathy.
9. History of significant valvular stenosis or regurgitation.
10. Patients with a pneumonectomy or more than moderate Chronic Obstructive Pulmonary Disease (COPD) or mild interstitial lung disease (ILD) or mild obstructive sleep apnea (OSA).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Incidence and Number of Adverse Events (AEs) | Up to 24 weeks
  An AE is any untoward medical occurrence in a patient or clinical trial patient administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. The incidence and number of patients who experience an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Monique Champagne, M.Sc, Study Director — 35Pharma Inc